CLINICAL TRIAL: NCT01439516
Title: Information and Financial Interventions for Kidney Donation in African Americans
Brief Title: Providing Resources to Enhance African American Patients' Readiness to Make Decisions About Kidney Disease (PREPARED) Study
Acronym: PREPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00011846; 1R01DK079682-01 (NIH)
Record Dates: First submitted 2011-08-31; First posted 2011-09-23 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: End Stage Renal Disease (ESRD); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Information (Experimental): Participants randomized to this arm of the study will received the PREPARED educational book and video.
  Interventions: Behavioral: Information
- Information and Financial Assistance (Experimental): Participants randomized to this arm of the study will receive the PREPARED educational book and video plus financial assistance for family members to cover costs associated with an evaluation for becoming a live kidney donor.
  Interventions: Behavioral: Information
- Usual Care (No Intervention): Participants randomized to this arm of the study will receive usual care from their physician.

INTERVENTIONS:
Behavioral: Information — Receipt of PREPARED educational book and video about treatments for end stage renal disease (ESRD)
  Arms: Information; Information and Financial Assistance

SUMMARY:
African Americans are less likely than Whites to receive kidney transplants, despite their being more than two-fold as likely as Whites to develop end stage renal disease (ESRD). Living related kidney donation (LD) offers patients an opportunity to bypass many barriers to receipt of deceased kidney transplants (e.g. waiting lists and immunological incompatibility), but minorities are less likely to receive living related kidney transplants (LRT). Evidence suggests African Americans may not discuss LD/LRT with their families or physicians at optimal rates, and thus may not have adequate information to initiate or participate in shared decision-making regarding LD/LRT. African Americans may also have financial concerns regarding convalescence and out of pocket expenses related to LD/LRT, another barrier impeding LD/LRT.

The primary goals of this study are to overcome these important barriers by enhancing ethnic minorities' consideration of LD/LRT through the promotion of shared decision-making regarding LD/LRT and provision of financial assistance for out of pocket expenses. The investigators specific aims are: a) to develop culturally sensitive informational (audiovisual) and financial interventions and b) to perform a randomized controlled trial to assess their effectiveness in increasing pursuit of LD/LRT among African American patients with ESRD and their families. The investigators hypothesize: (1) Patients and families who view informational materials designed to promote shared decision-making regarding LD/LRT will be more likely than patients and families not viewing these materials to discuss LD/LRT with family and with health care professionals. Patients and families viewing such informational materials will also be more likely than those not viewing these materials to pursue and complete the LD/LRT process and (2) patients and their families who are offered the intervention to promote shared decision-making plus a financial assistance intervention for potential live kidney donors will be more likely than patients and families not offered both interventions to pursue and complete the LD/LRT process.

DETAILED DESCRIPTION:
The investigators will enroll 210 adult African American patients with new-onset ESRD from dialysis facilities in the Baltimore metropolitan area and measure their initial commitment to pursue LD/LRT. Participants will then be randomized to one of three groups: 1) informational intervention alone (PREPARED education), 2) informational intervention plus living donor financial assistance program (PREPARED plus financial assistance), and 3) no intervention (Usual Care). The investigators will follow participants for up to 6 months for progression in their commitment to LD/LRT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* End-stage renal disease (ESRD) receiving hemodialysis for less than 2 years
* Self-reported as African-American
* English Speaking

Exclusion Criteria:

* Dementia
* Prior Kidney Transplant
* Non-English Speaking
* Cancer within 2 years prior to recruitment date
* Stage 4 Congestive Heart Failure
* End Stage Liver Disease
* Unstable Coronary Artery Disease
* Pulmonary Hypertension
* Severe Peripheral Vascular Disease
* Chronic Debilitating Infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pursuit of Living Related Transplantation | 6 months
  Measurement of patients' pursuit of LRT will be performed using a series of questions that assess the participants' knowledge, interest, and perceived barriers to LRT. We will also ascertain use of the living donor financial assistance among potential donors and completion of evaluation and kidney transplant among both patient participants and potential living donors.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Ebony Boulware, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Boulware LE, Ephraim PL, Ameling J, Lewis-Boyer L, Rabb H, Greer RC, Crews DC, Jaar BG, Auguste P, Purnell TS, Lamprea-Monteleagre JA, Olufade T, Gimenez L, Cook C, Campbell T, Woodall A, Ramamurthi H, Davenport CA, Choudhury KR, Weir MR, Hanes DS, Wang NY, Vilme H, Powe NR. Effectiveness of informational decision aids and a live donor financial assistance program on pursuit of live kidney transplants in African American hemodialysis patients. BMC Nephrol. 2018 May 3;19(1):107. doi: 10.1186/s12882-018-0901-x. PMID 29724177
- [Derived] Ephraim PL, Powe NR, Rabb H, Ameling J, Auguste P, Lewis-Boyer L, Greer RC, Crews DC, Purnell TS, Jaar BG, DePasquale N, Boulware LE. The providing resources to enhance African American patients' readiness to make decisions about kidney disease (PREPARED) study: protocol of a randomized controlled trial. BMC Nephrol. 2012 Oct 12;13:135. doi: 10.1186/1471-2369-13-135. PMID 23057616